CLINICAL TRIAL: NCT00867087
Title: An Open-label, Single-arm, Phase 2 Study Of Inotuzumab Ozogamicin Plus Rituximab In Subjects With Relapsed/Refractory Cd22-positive Diffuse Large B-cell Lymphoma, Eligible For Autologous Stem Cell Transplantation
Brief Title: Study Evaluating Inotuzumab Ozogamicin (CMC-544) Plus Rituximab In Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 3129K5-2005; B1931001 (Other: Alias Study Number); 2008-007802-12 (EudraCT Number)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2017-08-22 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma, B-Cell
Keywords: Diffuse large b-cell lymphoma; inotuzumab ozogamicin; autologous stem cell transplant
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Inotuzumab Ozogamicin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2 (Experimental): Inotuzumab ozogamicin, in combination with rituximab, will be administered to patients with relapsed/refractory diffuse large B-cell Non-Hodgkin's lymphoma prior to an autologous stem cell transplant (aSCT).
  Interventions: Drug: inotuzumab ozogamicin (CMC-544); Drug: rituximab

INTERVENTIONS:
Drug: inotuzumab ozogamicin (CMC-544) — 1.8 mg/m^2 every 21 days by intravenous infusion, 3 to 6 doses
  Other Names: cmc-544
Drug: rituximab — 375 mg/m^2 two days before cycle 1 by intravenous infusion; 375 mg/m^2 every 21 days by intravenous infusion, 3 to 6 doses

SUMMARY:
The purpose of this study is to evaluate inotuzumab ozogamicin in combination with rituximab prior to an autologous stem cell transplant (aSCT) in patients with relapsed/refractory diffuse large B-cell Non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* CD20/CD22-positive diffuse large B-cell NHL that has relapsed after 1 or 2 prior therapies; one prior therapy must include anthracyclines and one must include rituximab in combination with chemotherapy
* Relapsed/disease progression within 12 months after start of prior therapy and/or secondary International Prognostic Index (sIPI) score greater than 1
* Eligible for autologous stem cell transplant (aSCT)

Exclusion Criteria:

* Prior allogeneic hematopoietic stem cell transplant
* Within 6 months prior to test article: autologous transplant, treatment with anti-CD22 antibodies, radio-immunotherapy
* Veno-occlusive disease or sinusoidal obstruction syndrome, chronic liver disease, systemic vasculitides, current or chronic hepatitis B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2009-06-08 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (33):
- United States (19):
  - Loyola University Medical Center, Foster G. McGraw Hospital and Satellites, Maywood, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center (JTCC) at Hackensack University Medical Center (HUMC), Hackensack, New Jersey
  - Hackensack University Medical CenteR, Hackensack, New Jersey
  - John Theurer Cancer Center, Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UT Southwestern University Hospital - St. Paul, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - The University of Texas, M. D. Anderson Cancer Center, Houston, Texas
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare System of, San Antonio, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Pharmaceutical Research Center, Madison, Wisconsin
- France (7):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - CHU Saint-Eloi, Montpellier
  - Hopital Saint Louis, Paris
  - Hopital Haut-Leveque, Pessac
  - CH Lyon Sud, Pierre-Bénite
  - Departement d'Hematologie et d'Oncologie-, Strasbourg
- Charite Campus Virchow-Kilinikum-, Berlin, Germany
- Singapore General Hospital, Singapore, Singapore
- South Korea (3):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Asan Medical Center, Seoul, Seoul/korea
  - Severance Hospital, Yonsei University Health System, Seoul
- United Kingdom (2):
  - Christie Hospital, Manchester
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3129K5-2005&StudyName=Study%20Evaluating%20Inotuzumab%20Ozogamicin%20%28CMC-544%29%20Plus%20%20Rituximab%20In%20Diffuse%20Large%20B-Cell%20Non-Hodgkin%27s%20Lymphoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2: Intravenous (IV) inotuzumab ozogamicin 1.8 milligrams per square meter (mg/m^2) given on Day 2 of a 21-day cycle in combination with IV rituximab 375 mg/m^2 given on Day -2 (Cycle 1 only) and Day 1 as an induction therapy for a planned minimum of 3 cycles and a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Started | 63
Completed | 21
Not Completed | 42
Not completed — Other | 1
Not completed — Withdrawal by Subject | 4
Not completed — Death | 37

BASELINE CHARACTERISTICS:
Population: Safety population - included participants who received at least 1 dose of study medication (rituximab or inotuzumab ozogamicin).
Groups:
- Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2: IV inotuzumab ozogamicin 1.8 mg/m^2 given on Day 2 of a 21-day cycle in combination with IV rituximab 375 mg/m^2 given on Day -2 (Cycle 1 only) and Day 1 as an induction therapy for a planned minimum of 3 cycles and a maximum of 6 cycles.
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (12.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) After 3 Cycles of Inotuzumab Ozogamicin Plus Rituximab Therapy
Description: Response criteria based on National Cancer Institute (NCI) International Response Criteria for non-Hodgkin's lymphoma. CR: no detectable clinical & radiographic evidence of disease/disease-related symptoms; lymph nodes/nodal masses regressed to normal size (less than or equal to [≤] 1.5 cm in greatest transverse diameter for nodes greater than [>] 1.5 cm pre-therapy); spleen & other organs (if enlarged pre-therapy) regressed in size & spleen not palpable on physical examination; repeat bone marrow infiltrate clear. PR: > or equal to (≥) 50% decrease in sum of product diameters (SPD) of 6 largest dominant nodes/nodal masses; no increase in size of other nodes, liver, or spleen; splenic & hepatic nodules regressed by ≥ 50% in SPD; involvement of other organs usually assessable & no measurable disease present; no new sites of disease. Participants achieving CR, but with persistent morphologic bone marrow involvement or no bone marrow assessment after treatment were partial responders.
Time Frame: Up to 2 years (9 weeks of 3 21-day cycles and every 3 to 6 months during the long-term follow-up period)
Population: Intention-to-treat (ITT) population - included all participants enrolled into the study. Response includes confirmed CR/PR and unconfirmed CR/PR.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants | 28.6 [17.89 to 41.35]

2. Secondary Outcome: Kaplan-Meier Estimate of Progression Free Survival (PFS) 6 Months After Inotuzumab Ozogamicin Plus Rituximab Therapy
Description: PFS; time from date of randomization to earliest date of progression, relapse after CR, death from any cause without progression, start of new treatment for the lymphoma excluding treatments/procedures for consolidation therapy in this protocol, or censored at date of last tumor assessment. Progression: abnormal lymph nodes (long axis > 1.5 cm or long axis 1.1 to 1.5 cm and short axis > 1.0 cm); appearance of any new lesion > 1.5 cm in any axis during or at end of treatment; ≥ 50% increase from nadir in SPD of any previously involved nodes, in a single involved node, or in the size of other lesions; ≥ 50% increase in longest diameter of any single previously identified node > 1.0 cm in short axis.
Time Frame: 6 months after the first dose of inotuzumab ozogamicin
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants | 39.1 [26.9 to 51.1]

3. Secondary Outcome: Kaplan-Meier Estimate of PFS 2 Years After Inotuzumab Ozogamicin Plus Rituximab Therapy
Description: as for outcome 2
Time Frame: 2 years after the first dose of inotuzumab ozogamicin
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants | 25.3 [15.1 to 36.8]

4. Secondary Outcome: Percentage of Participants With a Response of CR or PR and Who Had Successful Granulocyte Colony Stimulating Factor (G-CSF) Mobilization of Peripheral Blood Stem Cells (PBSCs) Overall and After 3 Cycles of Inotuzumab Ozogamicin Plus Rituximab Therapy
Description: Successful mobilization of PBSC: ≥ 2 x 10^6 cluster of differentiation (CD) 34+ cells per kilogram (cells/kg) after 3 cycles. CR: no detectable clinical & radiographic evidence of disease/disease-related symptoms; lymph nodes/nodal masses regressed to normal size (≤ 1.5 cm in greatest transverse diameter for nodes > 1.5 cm pre-therapy); spleen & other organs (if enlarged pre-therapy) regressed in size & spleen not palpable on physical examination; repeat bone marrow infiltrate clear. PR: ≥ 50% decrease in SPD of 6 largest dominant nodes/nodal masses; no increase in size of other nodes, liver, or spleen; splenic & hepatic nodules regressed by ≥ 50% in SPD; involvement of other organs usually assessable & no measurable disease present; no new sites of disease. Participants achieving CR, but with persistent morphologic bone marrow involvement or no bone marrow assessment post treatment were partial responders. Response includes confirmed CR/PR and unconfirmed CR/PR.
Time Frame: From the first dose to approximately 2 to 3 weeks after 3 cycles of inotuzumab ozogamicin plus rituximab (induction) therapy (up to 12 weeks) and up to approximately 2 to 3 weeks after 6 cycles (up to 21 weeks).
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants
  Overall | 17.5 [9.05 to 29.10]
  After 3 cycles | 15.9 [7.88 to 27.26]

5. Secondary Outcome: Percentage of Participants With Successful G-CSF Mobilization of PBSC
Description: Successful mobilization of PBSC was defined as ≥ 2 x 10^6 CD34+ cells/kg collected after 3 cycles of inotuzumab ozogamicin plus rituximab therapy.
Time Frame: From the first dose to approximately 2 to 3 weeks after up to 6 cycles of inotuzumab ozogamicin plus rituximab (induction) therapy (up to 21 weeks).
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants | 28.6 [17.89 to 41.35]

6. Secondary Outcome: Percentage of Participants Who Underwent Autologous Stem Cell Transplant (aSCT)
Description: Participants underwent high dose chemotherapy and aSCT. In order to proceed to aSCT, participants were required to achieve CR or PR and successful collection of PSBC (≥ 2.0 x 10^6 CD34+ cells/kg collected after 3 cycles).
Time Frame: A minimum of 4 weeks and a maximum of 8 weeks after the last cycle of inotuzumab ozogamicin plus rituximab (induction) therapy (up to 26 weeks).
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants | 28.6 [17.89 to 41.35]

7. Secondary Outcome: Event-Free Survival (EFS) After aSCT
Description: EFS was the time (in months) from the date of aSCT to the earliest date of progression, relapse after CR, death from any cause without progression, initiation of a new treatment for the lymphoma or was censored at the date of the last tumor assessment.
Time Frame: From the completion of aSCT through 2 year long-term follow-up period, including but not limited to planned assessments scheduled every 3 to 6 months.
Population: ITT population. Only participants who underwent aSCT were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 18
Months | NA [4.1 to NA] — There were insufficient events to estimate the median and the upper bound of the 95% CI at the time of data analysis.

8. Secondary Outcome: Percentage of Participants With a CR After 3 Cycles of Inotuzumab Ozogamicin Plus Rituximab Therapy
Description: CR: complete disappearance of all detectable clinical & radiographic evidence of disease & disease-related symptoms; lymph nodes & nodal masses regressed to normal size (≤ 1.5 cm in their greatest transverse diameter for nodes > 1.5 cm before therapy); spleen and other organs (if enlarged prior to therapy) regressed in size & spleen not palpable on physical examination; repeat bone marrow infiltrate clear. Response includes confirmed CR and unconfirmed CR.
Time Frame: From the first dose to approximately 2 to 3 weeks after 3 cycles of inotuzumab ozogamicin plus rituximab (induction) therapy (up to 12 weeks).
Population: ITT population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants | 12.7 [5.65 to 23.50]

9. Secondary Outcome: Overall Survival (OS)
Description: OS was the time (in months) from the date of randomization to the date of death, and censored at the date of last contact if no death occurred.
Time Frame: From randomization until the date of death, or the date of last contact if no death occurred (up to 2 years).
Population: ITT population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Months | 12.5 [9.6 to NA] — Upper 95% CI could not be determined due to the pattern of censorship with respect to events.

10. Secondary Outcome: Percentage of Participants With Any Grade 3/4 Laboratory Abnormality During Therapy
Description: The following parameters were analyzed for serum chemistry; blood urea nitrogen (or urea), creatinine, glucose, calcium, sodium, potassium, phosphorus, lactate dehydrogenase, aspartate aminotransferase, alanine aminotransferase, total bilirubin (and direct bilirubin, if total bilirubin was elevated), alkaline phosphatase, uric acid (or urate), albumin and total protein. The following parameters were analyzed for hematology; lymphocytes, basophils, eosinophils, erythrocytes, hematocrit, hemoglobin, leukocytes, monocytes, neutrophils, platelets, prothrombin international normalized ratio, prothrombin time, fibrinogen, and activated partial thromboplastin time. Laboratory test results were graded using the NCI Common Terminology Criteria for Adverse Events, version 3.0 (CTCAE v3.0).
Time Frame: Within 3 days prior each dose of test article, on Day -2, 1, 8, and 15 of Cycles 1 to 3, 2 to 3 weeks after Cycle 3, at the end-of-treatment visit, and every 3 to 6 months during long-term follow-up (up to 2 years).
Population: Safety population
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants | 92.1

11. Secondary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) During Inotuzumab Ozogamicin Plus Rituximab Treatment
Description: An AE was any untoward, undesired, or unplanned event in the form of signs, symptoms, disease, or laboratory/physiologic observations occurring in a participant given a test article or in a clinical study; the event may not necessarily have had a causal relationship with the treatment. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; cancer. Treatment-emergent AEs were AEs that emerged after the first dose of the study treatment during the treatment period that were absent pre-treatment, or worsened during the treatment period relative to the pre-treatment state. The severity of all AEs was graded by the investigator using the NCI Common Terminology Criteria for AE Version 3.0 (CTCAE v3.0).
Time Frame: Treatment emergent AEs were collected from time of first dose to end of trial visit (participants not undergoing consolidation treatment) or until consolidation therapy. SAEs were collected from informed consent until end of trial visit (up to 6 months).
Population: Safety population Summary excludes events occurring after start of consolidation treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Number analyzed (Participants) | 63
Percentage of Participants
  Participants with AEs | 100.0
  Participants with SAEs | 34.9
  Participants with AEs Grade ≥ 3 | 90.5
  Participants with dose delayed due to AEs | 27.0
  Participants with dose reduced due to AEs | 11.1
  Participants permanently discontinued due to AEs | 9.5

ADVERSE EVENTS:
Time Frame: AEs collected from informed consent to end of treatment visit (participants not undergoing consolidation treatment) or until consolidation therapy. SAEs collected from informed consent until end of treatment visit for all participants (up to 6 months).
Description: The same event may appear as both an AE & SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant & non-serious in another, or 1 participant may have experienced both a serious & non-serious event during the study. Summaries inclusive of events occurring after start of consolidation treatment.
Arm/Group | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2
Serious Adverse Events (participants affected / at risk) | 29/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2 (N=63)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Aplasia (Congenital, familial and genetic disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
General physical health deterioration (General disorders) | 2
Multi-organ disorder (General disorders) | 1
Multi-organ failure (General disorders) | 1
Oedema (General disorders) | 1
Pyrexia (General disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 2
Bronchopneumonia (Infections and infestations) | 1
Candidiasis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Enterobacter infection (Infections and infestations) | 1
Enterobacter pneumonia (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Staphylococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Urinary tract infection enterococcal (Infections and infestations) | 1
Blood creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Encephalopathy (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 + Inotuzumab Ozogamicin 1.8 mg/m^2 (N=63)
Anaemia (Blood and lymphatic system disorders) | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 15
Lymphopenia (Blood and lymphatic system disorders) | 25
Neutropenia (Blood and lymphatic system disorders) | 22
Thrombocytopenia (Blood and lymphatic system disorders) | 43
Abdominal pain (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 18
Dyspepsia (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 32
Vomiting (Gastrointestinal disorders) | 16
Chills (General disorders) | 7
Fatigue (General disorders) | 26
Mucosal inflammation (General disorders) | 7
Oedema peripheral (General disorders) | 8
Pain (General disorders) | 6
Pyrexia (General disorders) | 21
Hyperbilirubinaemia (Hepatobiliary disorders) | 8
Upper respiratory tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 27
Blood alkaline phosphatase increased (Investigations) | 15
Blood lactate dehydrogenase increased (Investigations) | 7
Decreased appetite (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hypophosphataemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 14
Lethargy (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 4
Flushing (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less